CLINICAL TRIAL: NCT07312747
Title: Comparison Between Insertion of Bilateral Straight Cages Versus Unilateral Banana Cage in Lumbar Fusion Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Osman Ahmed Mahmoud, Resident at Neurosurgery Department, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: type of cages in lumbar fusion
Record Dates: First submitted 2025-11-21; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with bilateral straight cages (Active Comparator)
  Interventions: Procedure: cages in lumbar fusion surgery
- People with unilateral banana cage (Active Comparator)
  Interventions: Procedure: cages in lumbar fusion surgery

INTERVENTIONS:
Procedure: cages in lumbar fusion surgery — A critical factor in TLIF procedures is the type and positioning of the interbody cage. Traditionally, bilateral straight cages have been inserted to promote symmetrical load sharing and increase the surface area for fusion. This technique aims to ensure even support of the anterior column and reduce the risk of cage subsidence or pseudarthrosis. On the other hand, unilateral insertion of banana-shaped cages has been introduced as a potentially less invasive alternative that simplifies the procedure while still achieving adequate segmental stability and fusion

SUMMARY:
- To compare the clinical outcomes of bilateral straight cages and unilateral banana cage insertion in lumbar interbody fusion surgery, assess radiological outcomes, including intervertebral disc height, lumbar lordosis angle, and radiographic evidence of fusion, evaluate the rate of complications, such as cage migration, subsidence, pseudoarthrosis, and adjacent segment degeneration and analyze differences in operative time, blood loss, and length of hospital stay between the two techniques

DETAILED DESCRIPTION:
Lumbar fusion surgery is a widely utilized procedure for the treatment of a variety of spinal pathologies, including degenerative disc disease, lumbar spondylolisthesis, and spinal instability. Among the surgical techniques available, transforaminal lumbar interbody fusion (TLIF) has gained prominence due to its ability to access the disc space through a posterior approach, reduce neural retraction, and allow for thorough disc removal and interbody cage placement with minimal disruption to the spinal canal.(1)

A critical factor in TLIF procedures is the type and positioning of the interbody cage. Traditionally, bilateral straight cages have been inserted to promote symmetrical load sharing and increase the surface area for fusion. This technique aims to ensure even support of the anterior column and reduce the risk of cage subsidence or pseudarthrosis. On the other hand, unilateral insertion of banana-shaped cages has been introduced as a potentially less invasive alternative that simplifies the procedure while still achieving adequate segmental stability and fusion.(2,3) Despite growing adoption of both bilateral straight and unilateral banana cages, controversy remains regarding their relative biomechanical performance, clinical efficacy, and complication profiles. Factors such as asymmetrical load distribution in unilateral constructs, differences in cage surface area contact, and potential risks for adjacent segment degeneration or cage migration have yet to be definitively resolved through high-quality comparative studies.(4,5) This study protocol aims to compare the outcomes of bilateral straight cage versus unilateral banana cage insertion in lumbar spine fusion surgery. By evaluating parameters such as fusion rate, operative time, blood loss, cage subsidence, and patient-reported outcomes, the study will provide evidence-based insights to guide surgical technique selection and improve long-term outcomes for patients undergoing lumbar spine fusion surgery .(6,7)

ELIGIBILITY:
Inclusion Criteria:

* • Symptomatic discogenic low back pain with Radiological evidence of disc degeneration, instability, or spondylolisthesis

  * Failed medical treatment > 6 months

Exclusion Criteria:

* • Patients unfit for surgery .

  * Active spinal infection ,Osteoporosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
success rate of bilateral straight cages in lumbar fusion surgery | 6 months post operative
  Percentage of success of bilateral straight cages in lumbar fusion surgery
Percentage of success of unilateral banana cage in lumbar fusion surgery | 6 months Post operative

REFERENCES:
- [Result] Lang G, Perrech M, Navarro-Ramirez R, Hussain I, Pennicooke B, Maryam F, Avila MJ, Hartl R. Potential and Limitations of Neural Decompression in Extreme Lateral Interbody Fusion-A Systematic Review. World Neurosurg. 2017 May;101:99-113. doi: 10.1016/j.wneu.2017.01.080. Epub 2017 Jan 31. PMID 28153620
- [Result] Yoon J, Choi HY, Jo DJ. Comparison of Outcomes of Multi-Level Anterior, Oblique, Transforaminal Lumbar Interbody Fusion Surgery : Impact on Global Sagittal Alignment. J Korean Neurosurg Soc. 2023 Jan;66(1):33-43. doi: 10.3340/jkns.2022.0112. Epub 2022 Aug 23. PMID 35996945
- [Result] Della Pepa GM, La Rocca G, Barbagallo G, Spallone A, Visocchi M. Transient breathing disorders after posterior cervical surgery for degenerative diseases: pathophysiological interpretation. Eur Rev Med Pharmacol Sci. 2014;18(1 Suppl):89-92. PMID 24825050
- [Result] Ke W, Zhang T, Wang B, Hua W, Wang K, Cheung JPY, Yang C. Biomechanical Comparison of Different Surgical Approaches for the Treatment of Adjacent Segment Diseases after Primary Transforaminal Lumbar Interbody Fusion: A Finite Element Analysis. Orthop Surg. 2023 Oct;15(10):2701-2708. doi: 10.1111/os.13866. Epub 2023 Aug 24. PMID 37620961
- [Result] Malham GM, Ellis NJ, Parker RM, Seex KA. Clinical outcome and fusion rates after the first 30 extreme lateral interbody fusions. ScientificWorldJournal. 2012;2012:246989. doi: 10.1100/2012/246989. Epub 2012 Nov 1. PMID 23213282
- [Result] Drossopoulos PN, Ononogbu-Uche FC, Tabarestani TQ, Huang CC, Paturu M, Bardeesi A, Ray WZ, Shaffrey CI, Goodwin CR, Erickson M, Chi JH, Abd-El-Barr MM. Evolution of the Transforaminal Lumbar Interbody Fusion (TLIF): From Open to Percutaneous to Patient-Specific. J Clin Med. 2024 Apr 14;13(8):2271. doi: 10.3390/jcm13082271. PMID 38673544
- [Result] Daher M, Aoun M, El-Sett P, Kreichati G, Kharrat K, Sebaaly A. Unilateral Versus Bilateral Cages in Lumbar Interbody Fusions: A Meta-Analysis of Clinical and Radiographic Outcomes. World Neurosurg. 2024 Jun;186:158-164. doi: 10.1016/j.wneu.2024.03.142. Epub 2024 Mar 30. PMID 38561031